CLINICAL TRIAL: NCT04196140
Title: Evaluating the Safety and Effectiveness of the Omnipod Horizon™ Automated Glucose Control System in Patients With Type 1 Diabetes
Brief Title: Pivotal Omnipod Horizon™ Automated Glucose Control System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Horizon™ Pivotal Study
Record Dates: First submitted 2019-12-05; First posted 2019-12-12 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1D; Omnipod
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This is a single-arm, multi-center, prospective clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): All subjects wearing the Omnipod Horizon™ Automated Glucose Control System using the closed-loop algorithm.
  Interventions: Device: Omnipod Horizon™ Automated Glucose Control System

INTERVENTIONS:
Device: Omnipod Horizon™ Automated Glucose Control System — The Omnipod Horizon™ Automated Glucose Control System will provide automated insulin delivery

SUMMARY:
Subjects will undergo a 14-day outpatient, standard therapy phase during which sensor and insulin data will be collected. This will be followed by a 94-day (13-week) hybrid closed-loop phase conducted in an outpatient setting and an optional 12-month extension phase.

DETAILED DESCRIPTION:
The study schedule will consist of a standard therapy data collection phase followed by a hybrid closed-loop phase.

Subjects will undergo a 14-day outpatient, standard therapy phase (Phase 1 or ST) during which sensor and insulin data will be collected. Subjects, or their caregivers, will manage their diabetes at home per their usual routine using the study continuous glucose monitoring system (CGM) and remain on current multiple daily injections (MDI) or pump therapy. This will be followed by a 94-day (13-week) hybrid closed-loop phase (Phase 2), conducted in an outpatient setting where subjects, or their caregivers, will manage their diabetes at home using the Omnipod Horizon™ Automated Glucose Control System. After completing the 94-day hybrid closed-loop phase, subjects will have the option to continue using the system for an additional 12 months (Phase 3).

During the hybrid closed-loop phase, there will be supervised exercise challenges. A subset of subjects will participate in 5-days of supervised Meal and Exercise challenges. A subset of subjects will participate in 3-days of supervised HypoProtect Exercise challenges where comparisons were made between exercising in Automated Mode vs initiating HypoProtect 60 minutes prior to exercise vs initiating HypoProtect 30 minutes prior to exercise.

The hybrid closed-loop phase will begin on Study Day 1.

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent/assent 6-70 years
2. Subjects aged < 18 years must be living with parent/legal guardian
3. Diagnosed with type 1 diabetes for at least 6 months. Diagnosis is based on investigator's clinical judgment
4. Deemed appropriate for pump therapy per investigator's assessment taking into account previous history of severe hypoglycemic and hyperglycemic events, and other comorbidities
5. Investigator has confidence that the subject can successfully operate all study devices and is capable of adhering to the protocol
6. Willing to use only the following types of insulin during the study: Humalog, Novolog, Admelog or Apidra during the study
7. Must be willing to travel to and participate in meal and exercise challenges during 5-days of the hybrid closed-loop phase
8. Willing to wear the system continuously throughout the study
9. A1C <10% at screening visit
10. Must be willing to use the Dexcom App on the Omnipod Horizon™ Personal Diabetes Manager (PDM) as the sole source of Dexcom data (with the exception of the Dexcom Follow App) during the hybrid closed-loop phase
11. Subjects scoring ≥ 4 on the Clarke Questionnaire must agree to have an overnight companion, defined as someone who resides in the same home or building as the study subject and who can be available overnight
12. Able to read and speak English fluently
13. Willing and able to sign the Informed Consent Form (ICF) and/or has a parent/guardian willing and able to sign the ICF. Assent will be obtained from pediatric and adolescent subjects aged < 18 years per State requirements.

Exclusion Criteria:

1. A medical condition, which in the opinion of the investigator, would put the subject at an unacceptable safety risk
2. History of severe hypoglycemia in the past 6 months
3. History of DKA in the past 6 months, unrelated to an intercurrent illness, infusion set failure or initial diagnosis
4. Diagnosed with sickle cell disease
5. Diagnosed with hemophilia or any other bleeding disorders
6. Plans to receive blood transfusion over the course of the study
7. Currently diagnosed with anorexia nervosa or bulimia
8. Acute or chronic kidney disease (e.g. estimated GFR < 45) or currently on hemodialysis
9. History of adrenal insufficiency
10. Has taken oral or injectable steroids within the past 8-weeks or plans to take oral or injectable steroids during the course of the study
11. Unable to tolerate adhesive tape or has any unresolved skin condition in the area of sensor or pump placement
12. Plans to use insulin other than U-100 insulin intended for use in the study device during the course of the study
13. Use of non-insulin anti-diabetic medication other than metformin (e.g. GLP1 agonist, SGLT2 inhibitor, DPP-4 inhibitor, pramlintide)
14. Current or known history of coronary artery disease that is not stable with medical management, including unstable angina, or angina that prevents moderate exercise despite medical management, or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting within the previous 12-months.
15. For subjects >50 years old or with diabetes duration >20 years, abnormal electrocardiogram consistent with increased risk of arrhythmia, ischemia, or prolonged QTc interval (> 450 ms)
16. Thyroid Stimulating Hormone (TSH) is outside of normal range with clinical signs of hypothyroidism or hyperthyroidism
17. Pregnant or lactating, or is a woman of childbearing potential and not on acceptable form of birth control (acceptable includes abstinence, condoms, oral/injectable contraceptives, IUD or implant)
18. Participation in another clinical study using an investigational drug or device other than the Omnipod Horizon™ Automated Glucose Control System within the preceding 30-days or intends to participate during the study period
19. Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the investigator's clinical judgment

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Study Chair — Stanford University; Sue Brown, MD, Study Chair — University of Virginia
Locations (16):
- United States (16):
  - Stanford University, Palo Alto, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - University of Colorado Denver, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Atlanta Diabetes, Atlanta, Georgia
  - East Coast Institute for Research, Macon, Georgia
  - Northwestern University, Evanston, Illinois
  - Iowa Diabetes, West Des Moines, Iowa
  - Joslin Diabetes Center, Boston, Massachusetts
  - International Diabetes Center, Saint Louis Park, Minnesota
  - Mount Sinai, New York, New York
  - SUNY Syracuse, Syracuse, New York
  - University Hospitals Cleveland, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hood KK, Polonsky WH, MacLeish SA, Levy CJ, Forlenza GP, Criego AB, Buckingham BA, Bode BW, Hansen DW, Sherr JL, Brown SA, DeSalvo DJ, Mehta SN, Laffel LM, Bhargava A, Huyett LM, Vienneau TE, Ly TT. Psychosocial Outcomes with the Omnipod(R) 5 Automated Insulin Delivery System in Children and Adolescents with Type 1 Diabetes and Their Caregivers. Pediatr Diabetes. 2023 Jun 29;2023:8867625. doi: 10.1155/2023/8867625. eCollection 2023. PMID 40303234
- [Derived] Criego AB, Carlson AL, Brown SA, Forlenza GP, Bode BW, Levy CJ, Hansen DW, Hirsch IB, Bergenstal RM, Sherr JL, Mehta SN, Laffel LM, Shah VN, Bhargava A, Weinstock RS, MacLeish SA, DeSalvo DJ, Jones TC, Aleppo G, Buckingham BA, Ly TT. Two Years with a Tubeless Automated Insulin Delivery System: A Single-Arm Multicenter Trial in Children, Adolescents, and Adults with Type 1 Diabetes. Diabetes Technol Ther. 2024 Jan;26(1):11-23. doi: 10.1089/dia.2023.0364. Epub 2023 Nov 30. PMID 37850941
- [Derived] Hughes MS, Kingman RS, Hsu L, Lal RA, Buckingham BA, Zaharieva DP. Swimming With the Omnipod 5 Automated Insulin Delivery System: Connectivity in the Water. Diabetes Care. 2023 Aug 1;46(8):e148-e150. doi: 10.2337/dc23-0470. No abstract available. PMID 37311429
- [Derived] Polonsky WH, Hood KK, Levy CJ, MacLeish SA, Hirsch IB, Brown SA, Bode BW, Carlson AL, Shah VN, Weinstock RS, Bhargava A, Jones TC, Aleppo G, Mehta SN, Laffel LM, Forlenza GP, Sherr JL, Huyett LM, Vienneau TE, Ly TT; Omnipod 5 Research Group. How introduction of automated insulin delivery systems may influence psychosocial outcomes in adults with type 1 diabetes: Findings from the first investigation with the Omnipod(R) 5 System. Diabetes Res Clin Pract. 2022 Aug;190:109998. doi: 10.1016/j.diabres.2022.109998. Epub 2022 Jul 16. PMID 35853530
- [Derived] Brown SA, Forlenza GP, Bode BW, Pinsker JE, Levy CJ, Criego AB, Hansen DW, Hirsch IB, Carlson AL, Bergenstal RM, Sherr JL, Mehta SN, Laffel LM, Shah VN, Bhargava A, Weinstock RS, MacLeish SA, DeSalvo DJ, Jones TC, Aleppo G, Buckingham BA, Ly TT; Omnipod 5 Research Group. Multicenter Trial of a Tubeless, On-Body Automated Insulin Delivery System With Customizable Glycemic Targets in Pediatric and Adult Participants With Type 1 Diabetes. Diabetes Care. 2021 Jul;44(7):1630-1640. doi: 10.2337/dc21-0172. Epub 2021 Jun 7. PMID 34099518

RESULTS

PARTICIPANT FLOW:
Period: Phase 2
Arm/Group | Treatment
Started | 240
Completed | 235
Not Completed | 5
Period: Phase 3
Arm/Group | Treatment
Started | 224
Completed | 208
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138
  Male | 102
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 228
  Hispanic or Latino | 18
  Black or African American | 10
  Asian | 5
  Native Hawaiian or other Pacific Islander | 1
  American Indian or Alaskan Native | 4
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.8 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Severe Hypoglycemia (Events Per Person Months)
Description: Measure of serious device-related adverse events
Time Frame: Phase 2 hybrid closed-loop (94 days)
Measure: Number; unit: events per person month
Arm/Group | Treatment
Number analyzed (Participants) | 240
events per person month | .004

2. Primary Outcome: Incidence Rate of Diabetic Ketoacidosis (DKA) (Events Per Person Months)
Description: Measure of serious device-related adverse events
Time Frame: Phase 2 hybrid closed-loop (94 days)
Measure: Number; unit: events per person month
Arm/Group | Treatment
Number analyzed (Participants) | 240
events per person month | .001

3. Primary Outcome: Glycated Hemoglobin (A1C)
Description: Measures device effectiveness
Time Frame: 6 weeks continuous Phase 2 participation compared to baseline
Measure: Mean (Standard Deviation); unit: percentage of HbA1C
Arm/Group | Treatment
Number analyzed (Participants) | 240
percentage of HbA1C
  Baseline | 7.4 (0.9)
  Phase 2 | 6.9 (0.7)

4. Primary Outcome: Time in Range 70-180 mg/dL
Description: Measures device effectiveness
Time Frame: Phase 2 hybrid closed-loop (94 days) compared to Phase 1 standard therapy (14 days)
Measure: Mean (Standard Deviation); unit: % Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 240
% Time in Range
  Day Time ST | 58.6 (17.5)
  Day Time Phase 2 | 68.8 (10.7)
  Night Time ST | 60.1 (19.8)
  Night Time Phase 2 | 78.1 (12.6)
  Overall ST | 59.0 (17.2)
  Overall Phase 2 | 71.2 (10.2)

5. Secondary Outcome: Percent of Time >180 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: Phase 2 hybrid closed-loop (94 days) compared to Phase 1 standard therapy (14 days)
Measure: Mean (Standard Deviation); unit: % Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 240
% Time in Range
  Day Time ST | 39 (18.4)
  Day Time HCL | 29.5 (11)
  Night Time ST | 36.8 (20.7)
  Night Time HCL | 20.7 (12.6)
  Overall ST | 38.5 (18.1)
  Overall HCL | 27.3 (10.5)

6. Secondary Outcome: Percent of Time <70 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: Phase 2 hybrid closed-loop (94 days) compared to Phase 1 standard therapy (14 days)
Measure: Mean (Standard Deviation); unit: % Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 240
% Time in Range
  Day Time ST | 2.4 (2.78)
  Day Time HCL | 1.66 (1.38)
  Night Time ST | 3.11 (4.39)
  Night Time HCL | 1.17 (1.23)
  Overall ST | 2.57 (2.90)
  Overall HCL | 1.53 (1.25)

7. Secondary Outcome: Glycated Hemoglobin (A1C)
Description: Measures device effectiveness
Time Frame: at least 6 weeks and at least 8 weeks of continuous Phase 2 participation, end of Phase 2 (94 days), 6 months (180 days) and end of Phase 3 (270 days)
Measure: Mean (Standard Deviation); unit: % A1C
Arm/Group | Treatment
Number analyzed (Participants) | 240
% A1C
  6 Weeks Baseline | 7.4 (0.9)
  6 Weeks Phase 2 | 6.7 (0.6)
  8 Weeks Baseline | 7.4 (0.9)
  8 Weeks Phase 2 | 6.9 (0.7)
  6 months | 6.8 (0.6)
  12 months | 7.1 (0.7)

8. Secondary Outcome: Mean Glucose
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: Phase 2 hybrid closed-loop (94 days) and Phase 3 hybrid closed-loop (270 days) compared to Phase 1 standard therapy (14 days) during the day, overnight, and overall
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 240
mg/dL
  Day Time ST | 172.7 (32.2)
  Day Time Phase 2 | 159.4 (17.1)
  Day Time Phase 3 | 162.2 (19.7)
  Night Time ST | 167.8 (35.4)
  Night Time Phase 2 | 148.9 (19.2)
  Night Time Phase 3 | 150.8 (19.3)
  Overall ST | 171.5 (31.7)
  Overall Phase 2 | 156.7 (16.3)
  Overall Phase 3 | 159.3 (18.4)

9. Secondary Outcome: Percent of Time in Range 70-180 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: as for outcome 8
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 240
Percent Time in Range
  Day Time ST | 58.6 (17.5)
  Day Time Phase 2 | 68.8 (10.7)
  Day Time Phase 3: number analyzed (Participants) | 224
  Day Time Phase 3 | 67.0 (11.5)
  Night Time ST | 60.1 (19.8)
  Night Time Phase 2 | 78.1 (12.6)
  Night Time Phase 3: number analyzed (Participants) | 224
  Night Time Phase 3 | 76.6 (12.5)
  Overall ST | 59.0 (17.2)
  Overtime Phase 2 | 71.2 (10.2)
  Overtime Phase 3: number analyzed (Participants) | 224
  Overtime Phase 3 | 69.4 (10.8)

10. Secondary Outcome: Percent of Time in Range 70-140 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: as for outcome 8
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 240
Percent Time in Range
  Day Time ST | 36.0 (15.3)
  Day Time Phase 2 | 43.7 (10.6)
  Day Time Phase 3: number analyzed (Participants) | 224
  Day Time Phase 3 | 42.6 (11.1)
  Night Time ST | 38.2 (19.0)
  Night Time Phase 2 | 52.8 (15.5)
  Night Time Phase 3: number analyzed (Participants) | 224
  Night Time Phase 3 | 51.9 (14.4)
  Overall ST | 36.6 (15.4)
  Overall Phase 2 | 46.0 (10.7)
  Overall Phase 3: number analyzed (Participants) | 224
  Overall Phase 3 | 45.0 (10.8)

11. Secondary Outcome: Percent of Time >180 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: as for outcome 8
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 240
Percent Time in Range
  Day Time ST | 39.0 (18.4)
  Day Time Phase 2 | 29.5 (11.0)
  Day Time Phase 3: number analyzed (Participants) | 224
  Day Time Phase 3 | 31.3 (11.9)
  Night Time ST | 36.8 (20.7)
  Night Time Phase 2 | 20.7 (12.6)
  Night Time Phase 3: number analyzed (Participants) | 224
  Night Time Phase 3 | 22.0 (12.6)
  Overall ST | 38.5 (18.1)
  Overall Phase 2 | 27.3 (10.5)
  Overall Phase 3: number analyzed (Participants) | 224
  Overall Phase 3 | 28.9 (11.2)

12. Secondary Outcome: Percent of Time ≥ 250 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: as for outcome 8
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 240
Percent Time in Range
  Day Time ST | 14.7 (12.9)
  Day Time Phase 2 | 8.4 (6.3)
  Night Time ST | 13.2 (14.0)
  Night Time Phase 2 | 5.1 (6.2)
  Overall ST | 14.3 (12.5)
  Overall Phase 2 | 7.6 (5.8)
  Day Time Phase 3: number analyzed (Participants) | 224
  Day Time Phase 3 | 9.8 (7.4)
  Night Time Phase 3: number analyzed (Participants) | 224
  Night Time Phase 3 | 6.1 (6.1)
  Overall Phase 3: number analyzed (Participants) | 224
  Overall Phase 3 | 8.9 (6.7)

13. Secondary Outcome: Percent of Time ≥ 300 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: as for outcome 8
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 240
Percent Time in Range
  Day Time ST | 6.2 (7.9)
  Day Time Phase 2 | 2.8 (3.1)
  Day Time Phase 3: number analyzed (Participants) | 224
  Day Time Phase 3 | 3.7 (4.2)
  Night Time ST | 5.4 (8.6)
  Night Time Phase 2 | 1.7 (2.8)
  Night Time Phase 3: number analyzed (Participants) | 224
  Night Time Phase 3 | 2.2 (3.4)
  Overall ST | 6.0 (7.7)
  Overall Phase 2 | 2.5 (2.8)
  Overall Phase 3: number analyzed (Participants) | 224
  Overall Phase 3 | 3.3 (3.9)

14. Secondary Outcome: Percent of Time < 70 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: as for outcome 8
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 240
Percent Time in Range
  Day Time ST | 2.40 (2.78)
  Day Time Phase 2 | 1.66 (1.38)
  Day Time Phase 3: number analyzed (Participants) | 224
  Day Time Phase 3 | 1.75 (1.50)
  Night Time ST | 3.11 (4.39)
  Night Time Phase 2 | 1.17 (1.23)
  Night Time Phase 3: number analyzed (Participants) | 224
  Night Time Phase 3 | 1.38 (1.46)
  Overall ST | 2.57 (2.90)
  Overall Phase 2 | 1.53 (1.25)
  Overall Phase 3: number analyzed (Participants) | 224
  Overall Phase 3 | 1.66 (1.38)

15. Secondary Outcome: Percent of Time < 54 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: as for outcome 8
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 240
Percent Time in Range
  Day Time ST | 0.44 (0.99)
  Day Time Phase 2 | 0.29 (0.32)
  Day Time Phase 3 | 0.33 (0.38)
  Night Time ST | 0.77 (1.77)
  Night Time Phase 2 | 0.23 (0.35)
  Night Time Phase 3 | 0.34 (0.51)
  Overall ST | 0.52 (1.07)
  Overall Phase 2 | 0.27 (0.30)
  Overall Phase 3 | 0.33 (0.37)

16. Secondary Outcome: Standard Deviation (of Glucose)
Description: Glucose metric from study continuous glucose monitoring system (CGM)-measured glucose variability with the standard deviation (SD)
Time Frame: as for outcome 8
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 240
mg/dL
  Day Time ST | 62.4 (15.2)
  Day Time Phase 2 | 55.5 (11.9)
  Day Time Phase 3 | 57.9 (13.3)
  Night Time ST | 58.3 (16.3)
  Night Time Phase 2 | 45.6 (12.8)
  Night Time Phase 3 | 49.0 (13.9)
  Overall ST | 62.3 (14.9)
  Overall Phase 2 | 53.9 (11.6)
  Overall Phase 3 | 56.5 (13.0)

17. Secondary Outcome: Percent Coefficient of Variation (of Glucose)
Description: Glucose metric from study continuous glucose monitoring system (CGM)- measured glucose variability with the coefficient of variation (CV). Calculated by dividing the standard deviation of CGM values by the mean CGM values in the observation period.
Time Frame: as for outcome 8
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: Percent coefficient of variation
Arm/Group | Treatment
Number analyzed (Participants) | 240
Percent coefficient of variation
  Day Time ST | 36.1 (5.7)
  Day Time Phase 2 | 34.6 (5.2)
  Day Time Phase 3: number analyzed (Participants) | 224
  Day Time Phase 3 | 35.4 (5.2)
  Night Time ST | 34.9 (7.5)
  Night Time Phase 2 | 30.3 (5.9)
  Night Time Phase 3: number analyzed (Participants) | 224
  Night Time Phase 3 | 32.1 (6.2)
  Overall ST | 36.3 (5.6)
  Overall Phase 2 | 34.2 (5.1)
  Overall Phase 3: number analyzed (Participants) | 224
  Overall Phase 3 | 35.2 (5.2)

18. Secondary Outcome: Percentage of Time in Hybrid Closed-loop as Proportion of Overall Device Usage Time
Description: Measure of system usage
Time Frame: Phase 2 hybrid closed-loop (94 days) and Phase 3 (270 days)
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: Percent time spent
Arm/Group | Treatment
Number analyzed (Participants) | 240
Percent time spent
  Phase 2 Automated Mode | 95 (5.2)
  Phase 2 Manual Mode | 4.2 (4.7)
  Phase 3 Automated Mode: number analyzed (Participants) | 224
  Phase 3 Automated Mode | 93.6 (7.7)
  Phase 3 Manual Mode: number analyzed (Participants) | 224
  Phase 3 Manual Mode | 4.9 (6.9)

19. Secondary Outcome: Percent Glucose Management Indicator (% GMI)
Description: Glucose Management Indicator (%) approximates the laboratory hemoglobin A1c (%) expected based on average glucose readings from continuous glucose monitors from the last 14 days or more. Percent GMI provides information to a person with diabetes with how well their glucose is controlled over an extended period of time. A low value is more desirable than a high value, with a value of <7% being ideal for most people with diabetes. The calculation for GMI is as follows: GMI (%) = 3.31 + 0.02392 x (mean glucose reading in mg/dL from the last 14 days or more).
Time Frame: Phase 2 hybrid closed-loop (94 days) and Phase 3 hybrid closed-loop (270 days) compared to the Phase 1 standard therapy (14 days)
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: Percent GMI
Arm/Group | Treatment
Number analyzed (Participants) | 240
Percent GMI
  Day Time ST | 7.44 (0.77)
  Day Time Phase 2 | 7.12 (0.41)
  Day Time Phase 3: number analyzed (Participants) | 224
  Day Time Phase 3 | 7.19 (0.47)
  Night Time ST | 7.32 (0.85)
  Night Time Phase 2 | 6.87 (0.46)
  Night Time Phase 3: number analyzed (Participants) | 224
  Night Time Phase 3 | 6.92 (0.46)
  Overall ST | 7.41 (0.76)
  Overall Phase 2 | 7.06 (0.39)
  Overall Phase 3: number analyzed (Participants) | 224
  Overall Phase 3 | 7.12 (0.44)

20. Secondary Outcome: Total Daily Insulin (TDI) (Units)
Description: Measure of insulin requirements
Time Frame: as for outcome 19
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: units of insulin
Arm/Group | Treatment
Number analyzed (Participants) | 240
units of insulin
  ST | 41.7 (20.6)
  Phase 2 | 42.1 (19.3)
  Phase 3: number analyzed (Participants) | 224
  Phase 3 | 46.3 (20.1)

21. Secondary Outcome: Total Daily Insulin (TDI) (Units/kg)
Description: Measure of insulin requirements
Time Frame: as for outcome 19
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: units of insulin/kg
Arm/Group | Treatment
Number analyzed (Participants) | 240
units of insulin/kg
  ST | 0.72 (0.26)
  Phase 2 | 0.75 (0.28)
  Phase 3: number analyzed (Participants) | 224
  Phase 3 | 0.81 (0.32)

22. Secondary Outcome: Total Daily Basal Insulin (Units)
Description: Measure of insulin requirements
Time Frame: as for outcome 19
Population: 240 subjects were analyzed in Phase 2. 224 subjects were analyzed in Phase 3.
Measure: Mean (Standard Deviation); unit: units of insulin
Arm/Group | Treatment
Number analyzed (Participants) | 240
units of insulin
  ST | 19.7 (10.7)
  Phase 2 | 21.4 (10.5)
  Phase 3: number analyzed (Participants) | 224
  Phase 3 | 24.3 (10.8)

23. Secondary Outcome: Total Daily Basal Insulin (Units/kg)
Description: Measure of insulin requirements
Time Frame: as for outcome 19
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: units of insulin/kg
Arm/Group | Treatment
Number analyzed (Participants) | 240
units of insulin/kg
  ST | 0.33 (0.12)
  Phase 2 | 0.38 (0.15)
  Phase 3: number analyzed (Participants) | 224
  Phase 3 | 0.43 (0.18)

24. Secondary Outcome: Total Daily Bolus Insulin (Units)
Description: Measure of insulin requirements
Time Frame: as for outcome 19
Population: 240 subjects were analyzed in Phase 2. 224 subjects were analyzed in Phase 3.
Measure: Mean (Standard Deviation); unit: units of insulin
Arm/Group | Treatment
Number analyzed (Participants) | 240
units of insulin
  ST | 21.8 (12.7)
  Phase 2 | 20.7 (10.1)
  Phase 3: number analyzed (Participants) | 224
  Phase 3 | 22.0 (10.9)

25. Secondary Outcome: Total Daily Bolus Insulin (Units/kg)
Description: Measure of insulin requirements
Time Frame: as for outcome 19
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: units of insulin/kg
Arm/Group | Treatment
Number analyzed (Participants) | 240
units of insulin/kg
  ST | 0.39 (0.19)
  Phase 2 | 0.37 (0.15)
  Phase 3: number analyzed (Participants) | 224
  Phase 3 | 0.38 (0.17)

26. Secondary Outcome: Body Mass Index (BMI) (kg/m^2)
Description: Measure of change in weight
Time Frame: Phase 2 hybrid closed-loop (94 days) and Phase 3 hybrid closed-loop (270 days) compared to baseline
Population: 240 subjects were analyzed for Phase 2. 224 subjects were analyzed for Phase 3.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Treatment
Number analyzed (Participants) | 240
kg/m^2
  Baseline | 22.8 (5.7)
  Phase 2 | 23.0 (5.5)
  Phase 3 | 23.8 (5.6)

27. Other Pre Specified Outcome: Incidence Rate of Hypoglycemia (<70 mg/dL Confirmed by BG)
Description: Measure of device safety
Time Frame: HypoProtect compared to standard Omnipod 5 system use (3-day exercise challenge)
Measure: Number; unit: Percentage with hypoglycemia events
Arm/Group | Treatment
Number analyzed (Participants) | 50
Percentage with hypoglycemia events
  Exercise in Automated Mode without use of HypoProtect. | 40.8
  Hpt-60 (HypoProtect started 60 min before exercise.) | 34.7
  HPt-30 (HypoProtect started 30 min before exercise.) | 36.0

28. Other Pre Specified Outcome: Number of Hypoglycemic Events (<70 mg/dL Confirmed by BG)
Description: Number of hypoglycemic events less than 70mg/dL which was confirmed with a blood glucose reading.
Time Frame: HypoProtect compared to Automated Mode (3-day exercise challenge)
Measure: Number; unit: Number of events
Arm/Group | Treatment
Number analyzed (Participants) | 50
Number of events
  Automated Mode | 23
  HPt-60 | 19
  HPt-30 | 19

29. Other Pre Specified Outcome: Area Under the Curve (AUC) Less Than 70 mg/dL (Based on CGM Value)
Description: Measure of device effectiveness
Time Frame: HypoProtect compared to Automated Mode (3-day exercise challenge)
Measure: Mean (Standard Deviation); unit: hours x mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 50
hours x mg/dL
  Automated Mode | 58.3 (144.7)
  HPt-60 | 34.0 (83.9)
  HPt-30 | 34.3 (77.6)

30. Other Pre Specified Outcome: Minimum Continuous Glucose Monitor Value (Nadir Glucose)
Description: Measure of device effectiveness
Time Frame: HypoProtect compared to Automated Mode (3-day exercise challenge)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 50
mg/dL
  Automated Mode | 83.9 (25.0)
  HPt-60 | 94.9 (33.1)
  HPt-30 | 93.8 (32.8)

31. Other Pre Specified Outcome: Area Under the Curve (AUC) Greater Than 180 mg/dL (Based on CGM Value)
Description: Measure of device effectiveness
Time Frame: HypoProtect compared to Automated Mode (3-day exercise challenge)
Measure: Mean (Standard Deviation); unit: hours x mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 50
hours x mg/dL
  Automated Mode | 66.7 (243.4)
  HPt-60 | 30.0 (113.0)
  HPt-30 | 82.8 (400.7)

32. Other Pre Specified Outcome: Mean Absolute Decrease in Glucose (Based on CGM Value, From Start of Exercise to Nadir Glucose)
Description: Measure of device effectiveness
Time Frame: HypoProtect compared to Automated Mode (3-day exercise challenge)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 50
mg/dL
  Automated Mode | 58.1 (35.0)
  HPt-60 | 47.8 (35.6)
  HPt-30 | 42.0 (37.2)

33. Other Pre Specified Outcome: Carbohydrates Consumed During Exercise (Grams)
Description: Measure of device effectiveness
Time Frame: HypoProtect compared to Automated Mode (3-day exercise challenge)
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Treatment
Number analyzed (Participants) | 50
grams
  Automated Mode | 12.0 (15.5)
  HPt-60 | 10.1 (14.2)
  HPt-30 | 8.8 (12.3)

34. Other Pre Specified Outcome: Mean Glucose
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: Automated Mode compared to HypoProtect use during 70-minute exercise session and at 4-, 12-, and 24-hours post-exercise
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 50
mg/dL
  During Exercise Automated Mode | 117.6 (20.7)
  During Exercise HPt-60 | 123.2 (26.9)
  During Exercise HPt-30 | 119.7 (28.9)
  End of exercise through 4 hours post exercise Automated Mode | 150.6 (39.7)
  End of exercise through 4 hours post exercise HPt-60 | 156.9 (34.5)
  End of exercise through 4 hours post exercise HPt-30 | 167.2 (45.8)
  End of exercise through 12 hours post exercise Automated Mode | 156.7 (34.5)
  End of exercise through 12 hours post exercise HPt-60 | 153.6 (28.4)
  End of exercise through 12 hours post exercise HPt-30 | 155.2 (36.2)
  End of exercise through 24 hours post exercise Automated Mode | 150.8 (25.7)
  End of exercise through 24 hours post exercise HPt-60 | 150.0 (24.1)
  End of exercise through 24 hours post exercise HPt-30 | 151.4 (26.3)

35. Other Pre Specified Outcome: Percent of Time in Range 70-180 mg/dL
Description: Measure of device effectiveness
Time Frame: Automated Mode compared to HypoProtect use during 70-minute exercise session and at 4-, 12-, and 24-hours post-exercise
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Treatment
Number analyzed (Participants) | 50
Percent of time
  During Exercise Automated Mode | 88.9 (16.4)
  During Exercise HPt-60 | 90.4 (14.3)
  During Exercise HPt-30 | 89.5 (20.8)
  4-Hours Post Exercise Automated Mode | 69.4 (26.9)
  4-Hours Post Exercise HPt-60 | 66.9 (24.8)
  4-Hours Post Exercise HPt-30 | 66.6 (27.6)
  12 hours Post Exercise Automated Mode | 67.3 (23.8)
  12 Hours Post Exercise HPt-60 | 70.1 (20.2)
  12 Hours Post Exercise HPt-30 | 71.3 (22.1)
  24 Hours Post Exercise Automated Mode | 74.2 (17.1)
  24 Hours Post Exercise HPt-60 | 74.7 (17.1)
  24 Hours Post Exercise HPt-30 | 75.1 (16.6)

36. Other Pre Specified Outcome: Percent of Time > 180 mg/dL
Description: Measure of device effectiveness
Time Frame: Automated Mode compared to HypoProtect use during 70-minute exercise session and at 4-, 12-, and 24-hours post-exercise
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Treatment
Number analyzed (Participants) | 50
Percent of time
  During Exercise Automated Mode | 4.5 (11.4)
  During Exercise HPt-60 | 4.5 (13.0)
  During Exercise HPt-30 | 4.6 (18.6)
  4 Hours Post Exercise Automated Mode | 27.9 (28.0)
  4 Hours Post Exercise HPt-60 | 30.9 (25.9)
  4 Hours Post Exercise HPt-30 | 31.7 (28.0)
  12 Hours Post Exercise Automated Mode | 30.5 (24.1)
  12 Hours Post Exercise HPt-60 | 27.3 (19.9)
  12 Hours Post Exercise HPt-30 | 26.4 (22.9)
  24 Hours Post Exercise Automated Mode | 24.1 (17.5)
  24 Hours Post Exercise HPt-60 | 23.3 (16.9)
  24 Hours Post Exercise HPt-30 | 23.1 (16.9)

37. Other Pre Specified Outcome: Percent of Time ≥ 250 mg/dL
Description: Measure of device effectiveness
Time Frame: Automated Mode compared to HypoProtect use during 70-minute exercise session and at 4-, 12-, and 24-hours post-exercise
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Treatment
Number analyzed (Participants) | 50
Percent of time
  During Exercise Automated Mode | 0.3 (2.3)
  During Exercise HPt-60 | 0.0 (0.0)
  During Exercise HPt-30 | 0.0 (0.0)
  4 Hours Post Exercise Automated Mode | 6.3 (14.7)
  4 Hours Post Exercise HPt-60 | 4.5 (12.6)
  4 Hours Post Exercise HPt-30 | 12.0 (21.2)
  12 Hours Post Exercise Automated Mode | 7.0 (12.9)
  12 Hours Post Exercise HPt-60 | 7.1 (11.2)
  12 Hours Post Exercise HPt-30 | 8.4 (12.4)
  24 Hours Post Exercise Automated Mode | 5.3 (8.5)
  24 Hours Post Exercise HPt-60 | 5.8 (8.8)
  24 Hours Post Exercise HPt-30 | 7.0 (9.5)

38. Other Pre Specified Outcome: Percent of Time ≥ 300 mg/dL
Description: Measure of device effectiveness
Time Frame: Automated Mode compared to HypoProtect use during 70-minute exercise session and at 4-, 12-, and 24-hours post-exercise
Measure: Mean (Standard Deviation); unit: percent of time
Arm/Group | Treatment
Number analyzed (Participants) | 50
percent of time
  During Exercise Automated Mode | 0.0 (0.0)
  During Exercise HPt-60 | 0.0 (0.0)
  During Exercise HPt-30 | 0.0 (0.0)
  4 Hours Post Exercise Automated Mode | 1.4 (5.6)
  4 Hours Post Exercise HPt-60 | 1.8 (8.8)
  4 Hours Post Exercise HPt-30 | 5.3 (13.9)
  12 Hours Post Exercise Automated Mode | 2.4 (8.1)
  12 Hours Post Exercise HPt-60 | 2.5 (6.0)
  12 Hours Post Exercise HPt-30 | 3.3 (8.0)
  24 Hours Post Exercise Automated Mode | 1.6 (5.1)
  24 Hours Post Exercise HPt-60 | 1.7 (4.7)
  24 Hours Post Exercise HPt-30 | 2.2 (4.4)

39. Other Pre Specified Outcome: Percent of Time < 70 mg/dL
Description: Measure of device effectiveness
Time Frame: Automated Mode compared to HypoProtect use during 70-minute exercise session and at 4-, 12-, and 24-hours post-exercise
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Treatment
Number analyzed (Participants) | 50
Percent of time
  During Exercise Automated Mode | 6.52 (12.27)
  During Exercise HPt-60 | 5.12 (9.06)
  During Exercise HPt-30 | 5.88 (11.60)
  4 Hours Post Exercise Automated Mode | 2.72 (5.99)
  4 Hours Post Exercise HPt-60 | 2.17 (5.19)
  4 Hours Post Exercise HPt-30 | 1.68 (3.98)
  12 Hours Post Exercise Automated Mode | 2.21 (3.42)
  12 Hours Post Exercise HPt-60 | 2.65 (4.33)
  12 Hours Post Exercise HPt-30 | 2.33 (4.81)
  24 Hours Post Exercise Automated Mode | 1.72 (2.32)
  24 Hours Post Exercise HPt-60 | 2.00 (3.01)
  24 Hours Post Exercise HPt-30 | 1.78 (3.80)

40. Other Pre Specified Outcome: Percent of Time < 54 mg/dL
Description: Measure of device effectiveness
Time Frame: Automated Mode compared to HypoProtect use during 70-minute exercise session and at 4-, 12-, and 24-hours post-exercise
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Treatment
Number analyzed (Participants) | 50
Percent of time
  During Exercise Automated Mode | 1.40 (4.96)
  During Exercise HPT-60 | 0.52 (2.12)
  During Exercise HPT-30 | 0.37 (1.47)
  4 Hours Post Exercise Automated Mode | 0.38 (1.89)
  4 Hours Post Exercise HPt-60 | 0.60 (2.04)
  4 Hours Post Exercise HPt-30 | 0.26 (0.93)
  12 Hours Post Exercise Automated Mode | 0.40 (1.17)
  12 Hours Post Exercise HPt-60 | 0.62 (1.82)
  12 Hours Post Exercise HPt-30 | 0.70 (2.66)
  24 Hours Post Exercise Automated Mode | 0.26 (0.71)
  24 Hours Post Exercise HPt-60 | 0.41 (1.07)
  24 Hours Post Exercise HPt-30 | 0.44 (1.48)

41. Other Pre Specified Outcome: Standard Deviation (of Glucose)
Description: as for outcome 16
Time Frame: Automated Mode compared to HypoProtect use during 70-minute exercise session and at 4-, 12-, and 24-hours post-exercise
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 50
mg/dL
  During Exercise Automated Mode | 24.8 (13.8)
  During Exercise HPt-60 | 19.8 (11.6)
  During Exercise HPt-30 | 19.1 (11.3)
  4 Hours Post Exercise Automated Mode | 39.7 (17.7)
  4 Hours Post Exercise HPt-60 | 37.2 (16.1)
  4 Hours Post Exercise HPt-30 | 42.1 (24.2)
  12 Hours Post Exercise Automated Mode | 45.4 (19.0)
  12 Hours Post Exercise HPt-60 | 47.0 (20.0)
  12 Hours Post Exercise HPt-30 | 46.3 (19.0)
  24 Hours Post Exercise Automated Mode | 44.2 (15.3)
  24 Hours Post Exercise HPt-60 | 45.1 (17.5)
  24 Hours Post Exercise HPt-30 | 46.7 (16.2)

42. Other Pre Specified Outcome: Coefficient of Variation (of Glucose)
Description: Glucose metric from study continuous glucose monitoring system (CGM)-measured glucose variability with the coefficient of variation (CV). Calculated by dividing the standard deviation of CGM values by the mean CGM values in the observation period.
Time Frame: Automated Mode compared to HypoProtect use during 70-minute exercise session and at 4-, 12-, and 24-hours post-exercise
Measure: Mean (Standard Deviation); unit: Percent coefficient of variation
Arm/Group | Treatment
Number analyzed (Participants) | 50
Percent coefficient of variation
  During Exercise Automated Mode | 21.6 (11.7)
  During Exercise HPT-60 | 17.1 (10.4)
  During Exercise HPT-30 | 17.2 (11.2)
  4 Hours Post Exercise Automated Mode | 25.9 (8.5)
  4 Hours Post Exercise HPt-60 | 23.6 (8.4)
  4 Hours Post Exercise HPt-30 | 24.5 (10.7)
  12 Hours Post Exercise Automated Mode | 28.5 (8.1)
  12 Hours Post Exercise HPt-60 | 30.0 (9.8)
  12 Hours Post Exercise HPt-30 | 29.3 (8.6)
  24 Hours Post Exercise Automated Mode | 28.8 (6.3)
  24 Hours Post Exercise HPt-60 | 29.5 (8.6)
  24 Hours Post Exercise HPt-30 | 30.4 (7.5)

ADVERSE EVENTS:
Time Frame: Start of phase 2 (13 weeks) until the end of phase 3 (12 months).
Description: Adverse events listed below were collected during phase 2 and phase 3.
Groups:
- Phase 2: Subjects during the standard therapy phase (N=240) and phase 2 (N=240). During phase 2 subjects were using the Omnipod Horizon Automated Glucose Control System using the closed-loop algorithm.
- Phase 3: Subjects during phase 3 (N=224). During Phase 3 subjects were using the Omnipod Horizon Automated Glucose Control System using the closed-loop algorithm.
Arm/Group | Phase 2 | Phase 3
All-Cause Mortality (participants affected / at risk) | 0/240 | 1/224
Serious Adverse Events (participants affected / at risk) | 6/240 | 19/224
Other Adverse Events (participants affected / at risk) | 36/240 | 107/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2 (N=240) | Phase 3 (N=224)
Severe Hypoglycemia (Endocrine disorders) | 3 | 7
Diabetic Ketoacidosis (Endocrine disorders) | 1 | 1
Other (Investigations) | 2 | 9
Hypoglycemia (Endocrine disorders) | 0 | 1
Prolonged Hyperglycemia (Endocrine disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2 (N=240) | Phase 3 (N=224)
Hypoglycemia (Endocrine disorders) | 1 | 0
Prolonged Hyperglycemia (Endocrine disorders) | 18 | 40
Other (Investigations) | 14 | 58
Hyperglycemia (Endocrine disorders) | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT04196140/Prot_002.pdf
  • Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT04196140/SAP_001.pdf